CLINICAL TRIAL: NCT02839434
Title: Evaluation of the Interference of Antithrombotic Agents With Laboratory Monitoring of Heparin Therapy
Acronym: ACTARD
Status: Terminated | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AGR_2015_27
Record Dates: First submitted 2016-07-12; First posted 2016-07-21 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2017-09

CONDITIONS: Blood Coagulation Tests
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Treated with oral anticoagulants: Ex vivo study using blood samples from patients treated with oral anticoagulant (direct oral anticoagulants or AVK) at curative dose, taken in the usual cardiac monitoring.
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — This blood sample does not require specific puncture because it is made on the occasion of a sample justified by the patient monitoring.

SUMMARY:
Oral anticoagulants are increasingly prescribed and the are not discontinued for invasive cardiac procedures .

Additional parenteral anticoagulation is necessary for these procedures (FA ablation and invasive coronary explorations).

The unfractionated heparin doses are adapted on a monitoring test heparin, activated clotting time (ACT) with the aim of obtaining and maintaining an ACT > 300-400 sec. This goal is the same whether the patient is on oral anticoagulant treatment or not, and regardless of the initial level of anticoagulation.

The effects of oral anticoagulants on routine coagulation tests (PT, APTT, TT) are well documented, but few data have been published on the effects of heparin monitoring tests, particularly on the ACT.

The aim of this stuy is to redefine the target values of ACT and unfractionated heparin doses to administer to optimize the efficacy / safety of invasive procedures in cardiology.

ELIGIBILITY:
Inclusion Criteria:

* patient treated with oral anticoagulant at curative dose and requiring a requiring a venous blood sample for his management

Exclusion Criteria:

* opposition to the patient to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult treated with oral anticoagulant at curative dose
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Correlation between the plasmatic concentration in direct oral anticoagulants (DOAC) or International Normalized Ratio for AVK and the value of the Activated clotting time (ACT) | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation ophtalmique Adolphe de Rothschild, Paris, France